CLINICAL TRIAL: NCT00332644
Title: Pharmacotherapies: Efficacy, Mechanisms and Algorithms
Brief Title: Smoking Cessation Medications: Efficacy, Mechanisms and Algorithms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P50DA19706-1; P50DA019706 (NIH); NCT00109447 (obsolete NCT alias)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-10

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): nicotine patch alone treatment
  Interventions: Drug: nicotine patch
- 2 (Experimental): nicotine lozenge alone treatment
  Interventions: Drug: nicotine lozenge
- 3 (Experimental): nicotine patch + lozenge combination treatment
  Interventions: Drug: nicotine patch + nicotine lozenge
- 4 (Experimental): bupropion alone treatment
  Interventions: Drug: bupropion
- 5 (Experimental): bupropion + nicotine lozenge combination treatment
  Interventions: Drug: bupropion + lozenge
- 6 (Placebo Comparator): placebo control (no active medication) treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nicotine patch — used according to FDA package label
  Arms: 1
Drug: nicotine lozenge — used according to FDA-approved package directions
  Arms: 2
Drug: nicotine patch + nicotine lozenge — dosage of both according to FDA-approved dosing schedule
  Arms: 3
Drug: bupropion — dosage according to FDA-approved instructions
  Arms: 4
Drug: bupropion + lozenge — dosage according to FDA approved standard instructions
  Arms: 5
Drug: placebo — dosage same as active drug conditions
  Arms: 6

SUMMARY:
The proposed work will advance the understanding and effectiveness of tobacco dependence treatment and result in more smokers quitting successfully.

DETAILED DESCRIPTION:
This research study will last for three years. The first year involves a comparison of smoking cessation medications (bupropion, nicotine patch, and nicotine lozenge), including medications used in combination. The results of this study may allow researchers and clinicians to decide which medications are best for helping people to quit smoking as well as what treatments work best for different people. In addition, the first year of this study may help to clarify how these medications work.The purpose of the second and third years of this research study will be to get long-term results on the physical health, mental health, lifestyle factors, and the overall quality of life of people attempting to quit smoking. The results of this study may help researchers and clinicians better understand the health improvements that come from quitting or not quitting smoking.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 10 cigarettes per day for the previous 6 months - Expired CO > 9 ppm - Motivated to quit smoking - Able to read and write English - Willing to complete required study assessments

Exclusion Criteria:

* Uncontrolled hypertension (systolic >180mm Hg or diastolic >110mm Hg) - History of bipolar disorder or psychosis - Myocardial infarction or other serious cardiac problem in the previous 4 weeks - History of diagnosed anorexia and/or bulimia - Diagnosis of Alcohol Dependence in the previous 6 months by participant self-report or drinking 6 or more drinks on six or more days a week - History of seizure and/or serious head injury involving loss of consciousness - Use of contraindicated medications (MAO inhibitors, bupropion, lithium, anticonvulsants, antipsychotics) - Currently pregnant or breast-feeding - Unwilling to use effective contraception during the treatment phase - More than one participant from the same household - Allergic reactions to 3 or more classes of drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1504 (Actual)
Dates: Start 2004-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B. Baker, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW-CTRI Madison Research site, Madison, Wisconsin
  - UW-CTRI Milwaukee Research site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Burgess-Hull AJ, Roberts LJ, Piper ME, Baker TB. The social networks of smokers attempting to quit: An empirically derived and validated classification. Psychol Addict Behav. 2018 Feb;32(1):64-75. doi: 10.1037/adb0000336. Epub 2017 Dec 18. PMID 29251951
- [Derived] McCarthy DE, Ebssa L, Witkiewitz K, Shiffman S. Paths to tobacco abstinence: A repeated-measures latent class analysis. J Consult Clin Psychol. 2015 Aug;83(4):696-708. doi: 10.1037/ccp0000017. Epub 2015 Apr 13. PMID 25867447
- [Derived] Smith SS, Fiore MC, Baker TB. Smoking cessation in smokers who smoke menthol and non-menthol cigarettes. Addiction. 2014 Dec;109(12):2107-17. doi: 10.1111/add.12661. Epub 2014 Jul 21. PMID 24938369
- [Derived] Stein JH, Asthana A, Smith SS, Piper ME, Loh WY, Fiore MC, Baker TB. Smoking cessation and the risk of diabetes mellitus and impaired fasting glucose: three-year outcomes after a quit attempt. PLoS One. 2014 Jun 3;9(6):e98278. doi: 10.1371/journal.pone.0098278. eCollection 2014. PMID 24893290
- [Derived] Johnson HM, Piper ME, Baker TB, Fiore MC, Stein JH. Effects of smoking and cessation on subclinical arterial disease: a substudy of a randomized controlled trial. PLoS One. 2012;7(4):e35332. doi: 10.1371/journal.pone.0035332. Epub 2012 Apr 9. PMID 22496918
- [Derived] Asthana A, Piper ME, McBride PE, Ward A, Fiore MC, Baker TB, Stein JH. Long-term effects of smoking and smoking cessation on exercise stress testing: three-year outcomes from a randomized clinical trial. Am Heart J. 2012 Jan;163(1):81-87.e1. doi: 10.1016/j.ahj.2011.06.023. Epub 2011 Nov 14. PMID 22172440
- [Derived] Julius BR, Ward BA, Stein JH, McBride PE, Fiore MC, Colbert LH. Ambulatory activity associations with cardiovascular and metabolic risk factors in smokers. J Phys Act Health. 2011 Sep;8(7):994-1003. doi: 10.1123/jpah.8.7.994. PMID 21885891
- [Derived] Johnson HM, Gossett LK, Piper ME, Aeschlimann SE, Korcarz CE, Baker TB, Fiore MC, Stein JH. Effects of smoking and smoking cessation on endothelial function: 1-year outcomes from a randomized clinical trial. J Am Coll Cardiol. 2010 May 4;55(18):1988-95. doi: 10.1016/j.jacc.2010.03.002. Epub 2010 Mar 17. PMID 20236788
- See also: home page of agency performing the research — http://www.endcigs.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Patch: nicotine patch alone treatment for nicotine dependence.
- Nicotine Lozenge: nicotine lozenge alone treatment
- Nicotine Patch + Lozenge: nicotine patch + lozenge combination treatment
- Bupropion: bupropion alone treatment
- Bupropion + Nicotine Lozenge: bupropion + nicotine lozenge combination treatment
- Placebo Control: placebo control (no active medication) treatment
Period: Overall Study
Arm/Group | Nicotine Patch | Nicotine Lozenge | Nicotine Patch + Lozenge | Bupropion | Bupropion + Nicotine Lozenge | Placebo Control
Started | 262 | 260 | 267 | 264 | 262 | 189
Completed | 250 | 238 | 258 | 244 | 250 | 174
Not Completed | 12 | 22 | 9 | 20 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Patch | Nicotine Lozenge | Nicotine Patch + Lozenge | Bupropion | Bupropion + Nicotine Lozenge | Placebo Control | Total
Number analyzed (Participants) | 262 | 260 | 267 | 264 | 262 | 189 | 1504
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 252 | 256 | 262 | 256 | 256 | 179 | 1461
  >=65 years | 10 | 4 | 5 | 8 | 6 | 10 | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.6) | 45.3 (10.4) | 44.2 (11.1) | 43.9 (11.7) | 45.3 (10.4) | 43.1 (11.4) | 44.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 151 | 153 | 154 | 154 | 111 | 876
  Male | 109 | 109 | 114 | 110 | 108 | 78 | 628
Region of Enrollment [Number; unit: participants]
  United States | 262 | 260 | 267 | 264 | 262 | 189 | 1504

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence of Smoking, Biochemically (Exhaled CO) Confirmed
Description: Smoking status was assessed both as 7-day point-prevalence abstinence ("Have you smoked at all, even a puff, in the last 7 days?") and continuous abstinence (smoking at all since the target quit day), using a smoking calendar and the timeline follow-back method. All participants' self-reports of smoking status during study visits were confirmed by an expired carbon monoxide level of less than 10 ppm measured using a Micro-3 Smokerlyzer (Bedfont Scientific, Williamsburg, Virginia).
Time Frame: 6 months post quit date
Measure: Number; unit: participants with<10 ppm exhaled CO
Arm/Group | Nicotine Patch | Nicotine Lozenge | Nicotine Patch + Lozenge | Bupropion | Bupropion + Nicotine Lozenge | Placebo Control
Number analyzed (Participants) | 262 | 260 | 267 | 264 | 262 | 189
participants with<10 ppm exhaled CO | 90 | 87 | 107 | 84 | 87 | 42

ADVERSE EVENTS:
Time Frame: 6 months
Description: collection of data at all visits and phone contacts
Arm/Group | Nicotine Patch | Nicotine Lozenge | Nicotine Patch + Lozenge | Bupropion | Bupropion + Nicotine Lozenge | Placebo Control
Serious Adverse Events (participants affected / at risk) | 5/262 | 5/260 | 5/267 | 8/264 | 6/262 | 6/189
Other Adverse Events (participants affected / at risk) | 207/262 | 214/260 | 227/267 | 195/264 | 217/262 | 129/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch (N=262) | Nicotine Lozenge (N=260) | Nicotine Patch + Lozenge (N=267) | Bupropion (N=264) | Bupropion + Nicotine Lozenge (N=262) | Placebo Control (N=189)
hospitalization: cardiovascular (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
hospitalization: surgical (Surgical and medical procedures) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
hospitalization: respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Hopitalization: abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalization: psychiatric and alcohol (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Pregnancy
hospitalization: general (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death: COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch (N=262) | Nicotine Lozenge (N=260) | Nicotine Patch + Lozenge (N=267) | Bupropion (N=264) | Bupropion + Nicotine Lozenge (N=262) | Placebo Control (N=189)
cold (Infections and infestations) | 92 (92) | 102 (102) | 88 (88) | 74 (74) | 65 (65) | 57 (57)
cough (Infections and infestations) | 16 (16) | 13 (13) | 13 (13) | 9 (9) | 8 (8) | 7 (7)
dizziness (General disorders) | 7 (7) | 5 (5) | 9 (9) | 6 (6) | 15 (15) | 6 (6)
Dry mouth (General disorders) | 1 (1) | 0 (0) | 2 (2) | 20 (20) | 25 (25) | 3 (3)
flatulence (Gastrointestinal disorders) | 0 (0) | 10 (10) | 9 (9) | 0 (0) | 16 (16) | 4 (4)
flu (Infections and infestations) | 9 (9) | 16 (16) | 15 (15) | 7 (7) | 22 (22) | 10 (10)
headache (General disorders) | 26 (26) | 29 (29) | 34 (34) | 23 (23) | 30 (30) | 24 (24)
hiccups (General disorders) | 0 (0) | 35 (35) | 22 (22) | 0 (0) | 7 (7) | 1 (1)
heartburn (Gastrointestinal disorders) | 2 (2) | 31 (31) | 22 (22) | 2 (2) | 21 (21) | 1 (1)
nausea (Infections and infestations) | 25 (25) | 44 (44) | 55 (55) | 20 (20) | 33 (33) | 16 (16)
skin irritation (Skin and subcutaneous tissue disorders) | 85 (85) | 3 (3) | 63 (63) | 12 (12) | 15 (15) | 8 (8)
sleep disturbance (General disorders) | 67 (67) | 18 (18) | 63 (63) | 88 (88) | 69 (69) | 20 (20)
throat irritation (General disorders) | 7 (7) | 18 (18) | 21 (21) | 6 (6) | 16 (16) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No